CLINICAL TRIAL: NCT00675883
Title: COMPliance With Avonex® PS in Patients With Relapsing-Remitting MS
Acronym: COMPASS
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Vladimir Migounov, MD/Sr. Manager, Medical Affairs, Biogen Idec Canada Inc.
Other Study IDs: AVX-CAN-0703
Record Dates: First submitted 2008-05-08; First posted 2008-05-12 (Estimated); Last update posted 2012-01-30 (Estimated); Status verified 2012-01

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Prospective: 500 patients who will be enrolled in the MS Alliance program will be consented to participate in this study.
- Retrospective: 500 patient chart reviews will be completed for patients who were enrolled in the MS Alliance program between two (2) to three (3) years ago.

SUMMARY:
A phase IV, observational, survey-based study to measure compliance with Avonex® PS therapy in patients with Relapsing-Remitting Multiple Sclerosis, and to compare persistence on therapy 22 months after initial prescription of AVONEX® PS between patients enrolled in the current MS AllianceTM program versus patients enrolled in this program prior to October 2007.

DETAILED DESCRIPTION:
Study Design

Five hundred patients will be enrolled in the prospective portion of the study, all of whom will receive AVONEX. Patients will join the study by signing the attached Informed Consent Form (Appendix 1) at their doctor's office at the time of prescription. Innomar will provide the drug to approximately 40 new patients per month, so it will take about twelve to fourteen months to enroll all of the study subjects, assuming that all agree to participate. Once the recruitment period is over, it will take another 22 months to complete the study to the 22-months point for the last subject.

In the retrospective arm of the study, 500 chart reviews will be completed for patients who had participated in the MS Alliance program two (2) to three (3) years ago to determine persistence to therapy over a similar 22 month period.

Study Objectives

Primary Objectives:

- To assess patients' compliance (as defined above) with AVONEX therapy in the prospective arm using self-reported patients questionnaire, as well as to compare patients' persistence on therapy (as defined above) between prospective and retrospective arms.

Secondary Objective:

- Evaluate patients' satisfaction with new MSA program.

Patients and Methods

Only patients enrolled in the MSA program will be included in this study. There will be no interventions above the current standard of care with the MSA program. Two distinct patient arms will exist for this study: the prospective arm and the retrospective (chart review) arm.

Inclusion Criteria

* Diagnosed with Relapsing Remitting Multiple Sclerosis (RRMS)
* Prescription of AVONEX® PS (prefilled syringes)
* Enrolment in the MS AllianceTM program

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Relapsing Remitting Multiple Sclerosis (RRMS)
* Prescription of AVONEX® PS (prefilled syringes)
* Enrolment in the MS AllianceTM program

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled in the MS AllianceTM program
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2008-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Compliance with therapy in the prospective arm | Week 7-10 and Week 80-83
Persistence on therapy between prospective and retrospective arms | 22 months

SECONDARY OUTCOMES:
Patients' satisfaction with new MSA program | Week 7-10 and Week 80-83

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, London Health Sciences Centre, London, Ontario, Canada